CLINICAL TRIAL: NCT02730520
Title: Impact of Age on the Prevalence of Allergic Sensitization
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Olivier Michel, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-Age-Allergy
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Allergy
Keywords: respiratory disease; allergen sensitization; aging; skin tests; air allergens
MeSH Terms: conditions — Hypersensitivity; Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Immuno-allergology patients: Patients followed within the Immuno-Allergology Service of the CHU Brugmann Hospital, who received an allergy assessment between 01/01/2015 and 31/12/2015. At least 1400 dermis will be analyzed. The allergens tested include: dermatophagoides pteronyssinus (DEPT), dermatophagoides farinae (DPF), blomia, cat, dog, cockroach, orchardgrass, timothy grass, alder, hazel,birch, olive tree, cypress, ash, latex, aspergillus, alternaria, cladosporium, peanut, hazel.
  Interventions: Other: Retrospective analysis of patient files

INTERVENTIONS:
Other: Retrospective analysis of patient files — The results of the allergen skin tests will be encoded as the edema diameter. The allergenicity score (mean of the skin reactivities for each allergen) will be compared between each age groups. The impact of tabagism, gender, BMI and residential area on the allergic reactivity will also be assessed in the overall population and within each age group.

SUMMARY:
Worldwide, respiratory diseases have a significant impact on morbidity and mortality of individuals.Tobacco, lifestyle and certain allergens such as dust mites play an important role in the prevalence and morbidity of these diseases. Scientific literature indicates that sensitization to allergens and respiratory diseases (asthma, rhinitis, chronic obstructive pulmonary disease) are closely linked. Moreover, smoking has an effect on allergen sensitivity.

To make a diagnosis of allergic sensitization, skin tests are performed in the patient. One of the methods used is the technique of "prick test". In practice, a drop of purified allergen extract is placed on the patient's skin (arms or back). A little dosis of the product is then injected in the epidermis. If fifteen minutes later, there is an edematous reaction, its diameter is measured in millimeters. From 4 mm, it is considered that the patient is sensitized to the tested foods or allergens.This technique is painless and convenient to patients of all ages, including newborns or conversely very aged patients.

This is a retrospective study based on the encoding and statistical analysis of data collected in patients followed within the Immuno-Allergology Service of the CHU Brugmann Hospital, who received an allergy assessment between 01/01/2015 and 31/12/2015. The allergens tested include: dermatophagoides pteronyssinus (DEPT), dermatophagoides farinae (DPF), blomia, cat, dog, cockroach, orchardgrass, timothy grass, alder, hazel,birch, olive tree, cypress, ash, latex, aspergillus, alternaria, cladosporium, peanut, hazel.

At least 1400 files will be analyzed.

Patients will be distributed in six age groups.The results of the allergen skin tests will be encoded as the edema diameter. The allergenicity score (mean of the skin reactivities for each allergen) will be compared between each age groups. The impact of tabagism, gender, BMI and residential area on the allergic reactivity will also be assessed in the overall population and within each age group.

The main objective is to evaluate the effect of age on the skin test positivity. The secondary objective is to highlight the environmental factors that have an impact on allergic diseases.

ELIGIBILITY:
Inclusion Criteria:

* All patients followed within the Immuno-Allergology Service of the CHU Brugmann Hospital
* Who received an allergy assessment between 01/01/2015 and 31/12/2015. The allergens tested include: dermatophagoides pteronyssinus (DEPT), dermatophagoides farinae (DPF), blomia, cat, dog, cockroach, orchardgrass, timothy grass, alder, hazel,birch, olive tree, cypress, ash, latex, aspergillus, alternaria, cladosporium, peanut, hazel.

Exclusion Criteria:

* Negative histamine patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed within the Immuno-Allergology Service of the CHU Brugmann Hospital, who received an allergy assessment between 01/01/2015 and 31/12/2015.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Allergenicity score | one year (01/01/2015 to 31/12/2015)
  Mean of the skin reactivities for each allergen. The results of the allergen skin tests are encoded as the edema diameter. Scores will be compared between the different age groups.

SECONDARY OUTCOMES:
Smoking status | one year (01/01/2015 to 31/12/2015)
  Effect of the smoking/non smoking status on the allergic reactivity, analysed in the hole group and in the different age groups.
Geographic localisation | one year (01/01/2015 to 31/12/2015)
  Effect of the area of residence on the allergic reactivity, analysed in the hole group and in the different age groups.
Sex | one year (01/01/2015 to 31/12/2015)
  Gender effect on the allergic reactivity, analysed in the hole group and in the different age groups.
Body Mass Index | one year (01/01/2015 to 31/12/2015)
  Effect of the body mass index on the allergic reactivity, analysed in the hole group and in the different age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Michel, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Bauchau V, Durham SR. Epidemiological characterization of the intermittent and persistent types of allergic rhinitis. Allergy. 2005 Mar;60(3):350-3. doi: 10.1111/j.1398-9995.2005.00751.x. PMID 15679721